CLINICAL TRIAL: NCT06249334
Title: Whole-Body Electrical Stimulation in Patients Undergoing Lung Transplantation: Randomized Clinical Trial
Brief Title: Whole-Body Electrical Stimulation in Patients Undergoing Lung Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBES_LT
Record Dates: First submitted 2023-11-29; First posted 2024-02-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-02

CONDITIONS: Lung Transplantation; Electric Stimulation
Keywords: Lung transplantation; Electric stimulation; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole-body electrical stimulation (WB-EMS) (Experimental): WB-EMS will be performed with ReCare® equipment (Visuri, Minas Gerais, Brazil). Patients will perform sessions once a day, totaling a maximum of 15 sessions. In addition to the WB-EMS protocol, the patients will receive routine physiotherapy at the hospital.
  Interventions: Other: Whole-body electrical stimulation
- Routine physical therapy (Active Comparator): Patients in the control group (active comparator) will receive routine hospital physical therapy until the moment of hospital discharge.
  No intervention with electrical stimulation will be performed in this group.
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Whole-body electrical stimulation — The protocol with whole-body electrical stimulation will begin in the intensive care unit and will be completed in the inpatient unit. To stimulate all proposed muscle groups, self-adhesive electrodes will be positioned bilaterally on the quadriceps femoris, tibialis anterior, biceps brachii and lower rectus abdominis muscles. The frequency of 75 Hz will be adopted and the intensity will be adjusted to cause visible muscle contraction. The progression of the therapy protocol will occur throughout the sessions aiming to reach 20 minutes of therapy and 80 contractions.
  Other Names: Whole-body electromyostimulation
  Arms: Whole-body electrical stimulation (WB-EMS)
Other: Routine physical therapy — The protocol will be based on knee and hip flexion and extension movements; hip adduction and abduction; flexion and extension of shoulders, elbows and wrists; shoulder abduction and adduction; respecting the range of each joint. Volunteers will also perform transfers from lying to sitting and standing positions. Respiratory conduct will be based on ventilation patterns, bronchial hygiene maneuvers and cough.
  Arms: Routine physical therapy

SUMMARY:
This study aims to evaluate the effects of whole-body electrical stimulation (WB-EMS) in the rehabilitation of patients undergoing lung transplantation. This is a randomized clinical trial with patients from the inpatient unit of Dom Vicente Scherer Hospital of Irmandade Santa Casa de Misericórdia from Porto Alegre (ISCMPA) who will be allocated to a control group (which will receive physiotherapy from routine) or intervention group (which will receive physiotherapy from routine and WB-EMS). Interventions with WB-EMS will occur every day from the moment of extubation until hospital discharge (15 sessions per patient). Assessments will be carried out pre-lung transplantation, after extubation, during intervention protocols and at the time of hospital discharge.

DETAILED DESCRIPTION:
Patients on the lung transplant list may experience post-procedure complications that culminate in a higher risk of mortality, which are related to primary and chronic graft dysfunction and infections. These complications are partly responsible for prolonged immobility, sarcopenia, decline in functional capacity and deterioration in quality of life. There is evidence that physical rehabilitation, mainly through exercise, improves the physical capacity and quality of life of transplant patients. However, not all patients are able to perform this type of activity due to low tolerance for it. In this sense, WB-EMS can be an alternative for early rehabilitation. This study aims to evaluate the effects of WB-EMS in the rehabilitation of patients undergoing lung transplantation.

Patients will be selected from the Pulmonary Rehabilitation Center of Pereira Filho Hospital prior to lung transplantation and the following assessments will be carried out: muscle architecture and quality (ultrasound), peripheral muscle strength (dynamometry of lower and upper limbs, Medical Research Council scale and 10-repetition sit-and-stand test), respiratory muscle strength (manovacuometry) and functional capacity (six-minute walk test). After the transplant, with the patient admitted to the intensive care unit, and after being extubated, blood sample will be collected to measure muscle damage, also it will be evaluated the muscle architecture and quality, peripheral muscle strength (only using the Medical Research Council scale) and respiratory muscle strength. Prior to hospital discharge, muscle architecture and quality, peripheral muscle strength (dynamometry of lower and upper limbs, Medical Research Council scale and 10-repetition sit-and-stand test), respiratory muscle strength, functional capacity, and muscle damage will be reassessed, along with the length of hospital stay.

During the training period, the safety of the therapy will be assessed by monitoring cardiorespiratory parameters, muscle pain (analogic visual scale) and fatigue (Borg subjective perceived exertion scale).

Patients will be randomized to the control group (GC) (which will receive physiotherapy from routine) or the intervention group (GI), which will perform whole-body electrical stimulation using the equipment ReCARE® (Visuri, Minas Gerais, Brazil), in addition to routine physiotherapy. After extubation, patients will begin the protocol for 15 sessions and will be reevaluated, therefore the protocol begins in the intensive care unit and will be completed in the inpatient unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral or bilateral lung transplantation;
* Admitted to the intensive care unit and without invasive ventilatory support;
* Hemodynamically stable;
* Time less than or equal to 7 days between lung transplantation and the beginning of rehabilitation protocols.

Exclusion Criteria:

* Patients with severe psychomotor agitation;
* Recent acute myocardial infarction (24 hours) and / or uncontrolled arrhythmias;
* Temporary transcutaneous pacemaker;
* Stroke after lung transplantation;
* Decompensated heart failure;
* Uncontrolled hypertension (systolic blood pressure > 230 mmHg and diastolic blood pressure > 120 mmHg) or mean arterial pressure <60 mmHg;
* Patients who present important hemodynamic changes during training;
* Peripheral vascular changes in the lower limbs such as untreated deep vein thrombosis;
* In a feverish state;
* Patients with epidermal lesions on the thighs that make it impossible to place self-adhesive electrodes for electrical stimulation;
* Patients with acute renal failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Isometric quadriceps muscle strength. | Time 0 (baseline) and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Isometric quadriceps muscle strength will be evaluated using a portable dynamometer.
Lower limb muscle strength. | Time 0 (baseline) and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Lower limb strength will be carried out using the 10-repetition sit-and-stand test (SST).
Mortality. | Mortality will be assessed after 30 days, after 60 days and up to 1 year after lung transplantation.
  Mortality will be assessed by counting the number of deaths occurring in the study and after hospital discharge.

SECONDARY OUTCOMES:
Safety of whole-body electrical stimulation. | Time 0 (pre intervention), after 10 minutes and at 20 minutes from the beginning of the intervention.
  Safety of whole-body electrical stimulation will be assessed by measuring peripheral oxygen saturation.
Safety of whole-body electrical stimulation. | Time 0 (pre intervention), after 10 minutes and at 20 minutes from the beginning of the intervention.
  Safety of whole-body electrical stimulation will be assessed by measuring heart rate.
Safety of whole-body electrical stimulation. | Time 0 (pre intervention), after 10 minutes and at 20 minutes from the beginning of the intervention.
  Safety of whole-body electrical stimulation will be assessed by measuring blood pressure.
Muscle pain. | Time 0 (pre intervention), after 10 minutes and at 20 minutes from the beginning of the intervention.
  Muscle pain will be measured with the analogic visual scale (AVS). This scale classifies pain from 0 (not at all) to 10 (maximum).
Safety of whole-body electrical stimulation. | Time 0 (pre intervention), after 10 minutes and at 20 minutes from the beginning of the intervention.
  Safety of whole-body electrical stimulation will be assessed by perceived exertion with the modified Borg Scale.This scale classifies effort from 0 (nothing at all) to 10 (maximum).
Isometric muscle strength of the elbow flexors. | Time 0 (baseline) and immediately after 15 sessions (totaling a maximum of 3 weeks).
  The muscle strength of the upper limbs will be assessed through isometric contraction of the elbow flexor muscles with a portable dynamometer.
Upper limb muscle strength. | Time 0 (baseline) and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Palmar handgrip will also be assessed using an analog hydraulic dynamometer.
Overall muscle strength. | Time 0 (baseline), on the first day after extubation and immediately after 15 sessions (totaling a maximum of 3 weeks).
  To assess global muscle strength, the Medical Research Council (MRC) scale will be used. The total score ranges from 0 (quadriplegia) to 60 points (preserved muscle strength).
Respiratory muscle strength. | Time 0 (baseline), on the first day after extubation and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Respiratory muscle strength will be measured using the digital manovacuometer.
Muscle architecture. | Time 0 (baseline), on the first day after extubation and immediately after 15 sessions (totaling a maximum of 3 weeks).
  The muscle architecture will be evaluated for the acquisition of ultrasound images of the vastus lateralis, rectus femoris, biceps brachii and rectus abdominis muscles, using a high-resolution ultrasound.
Functional capacity. | Time 0 (baseline) and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Functional capacity will be assessed using the six-minute walk test (6MWT).
Muscle damage. | On the first day post extubation and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Muscle damage will be assessed by dosage of creatine phosphokinase.
Muscle damage. | On the first day post extubation and immediately after 15 sessions (totaling a maximum of 3 weeks).
  Muscle damage will be assessed by dosage of lactate dehydrogenase.
Length of hospital stay. | From randomization to discharge or death from any cause, whichever comes first, assessed up to 3 months.
  Length of hospital stay will be based on the number of days between the date of admission and hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jociane Schardong, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande Do Sul (RS), Brazil

REFERENCES:
- [Derived] Garlet AB, Plentz RDM, Righi NC, Schardong J. Whole-body electrical stimulation in patients undergoing lung transplantation in Southern Brazil: study protocol of a single-center randomized controlled trial. Trials. 2025 Dec 5;27(1):23. doi: 10.1186/s13063-025-09177-y. PMID 41350869